CLINICAL TRIAL: NCT01432574
Title: A Phase II Study of Gardasil in Human Papillomavirus Research The Mid-Adult Male Vaccine Study - The MAM STUDY
Brief Title: Study of Gardasil in Mid-Adult Males (MAM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-16593
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Human Papillomavirus
Keywords: HPV
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Papillomavirus Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gardasil Vaccine (Experimental): Vaccine Administration: A total of 3 injections (shots) at 3 separate visits.
  Interventions: Biological: Gardasil

INTERVENTIONS:
Biological: Gardasil — The First Shot: Given on the day participants joined the study (Visit 1). The Second Shot: Given about 2 months later (Visit 2). The Third Shot: Given about 6 months after the first (Visit 3).
  Other Names: HPV vaccine

SUMMARY:
The purpose of this study is to test the effectiveness of the research study vaccine, Gardasil, in men ages 27-45 who have completed 4 years of observation in The Human Papillomavirus [HPV] infection in men (HIM) Study.

DETAILED DESCRIPTION:
The MAM Study is a prospective pilot intervention trial to investigate patterns of human papillomavirus (HPV) vaccine immunogenicity in men, aged 27-45 years, in which the men will receive Gardasil. Gardasil was administered at 0, 2, and 6 months. Blood was drawn at 0 and 7 months to provide a quadrivalent HPV antibody serologic profile. Participants also completed surveys via computer-assisted interviews (CASI) at Day 1 and Month 7 to record sexual behavior.

Our overall goal is to test the efficacy of Gardasil to reduce HPV 6, 11, 16, 18 persistent infection among men at the external genital epithelium, anal canal, and oral cavity, and to reduce lesions caused by these HPV types at the external genital epithelium and anal canal. The purpose of this Phase II trial is to establish the immunogenicity of Gardasil among mid-adult men and to establish the infrastructure with which to build the larger Phase III trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Men that have completed 4 years of follow-up in the on-going international prospective natural history study of HPV in men (The HIM Study)
* Willing to comply with 4 scheduled visits within a 7-month period

Exclusion Criteria:

* Have received an HPV vaccine
* Have a prior diagnosis of penile or anal cancers
* Have a prior diagnosis of high grade anal intraepithelial neoplasia
* Have been diagnosed with human immunodeficiency virus (HIV)/acquired immune deficiency syndrome (AIDS)
* Have a history of anaphylaxis to vaccines
* Have known impairment of the immune system
* Have received any blood products within 6 months of enrollment

Ages: 27 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-02-19 (Actual); Primary Completion 2014-05-23 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Giuliano, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (2):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States
- National Institute of Public Health, Mexico, Cuernavaca, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIM Study participants that met the eligibility criteria were invited and enrolled into this Phase II Trial at the US and Mexico clinical sites between February and October of 2013.
Period: Overall Study
Arm/Group | Gardasil Vaccine
Started | 150
Completed | 147
Not Completed | 3
Not completed — Moved | 2
Not completed — Not interested | 1

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Gardasil Vaccine
Number analyzed (Participants) | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 150
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 36 [27 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 150
Race/Ethnicity, Customized [Number; unit: participants]
  White | 68
  Black/African American | 12
  Asian/Pacific Islander | 3
  Native American/Alaskan | 1
  More than one race | 65
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 75
  Mexico | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Seropositive at Month 7
Description: Immune response was measured with a multiplex competitive Luminex immunoassay (anti-HPV-6, -11, -16, and -18 chemiluminescence immunoassay analyzer (cLIA); Merck) at Pharmaceutical Product Development (PPD). Briefly, this assay simultaneously quantitates neutralizing antibodies to HPV 6, 11, 16, and 18 in 50 μL of serum. The seronegative study population at Day 1 (no detectable HPV antibody titers at Day 1) were to be categorized as seroconverted due to increase in titer levels for each vaccine component at Month 7.
Time Frame: 7 Months
Population: Participants who had specimens contributing to both Day 1 and Month 7 serum HPV antibody evaluations.
Measure: Number; unit: percentage of participants
Arm/Group | Gardasil Vaccine - Month 7
Number analyzed (Participants) | 145
percentage of participants
  HPV 6 | 100
  HPV 11 | 100
  HPV 16 | 100
  HPV 18 | 100

2. Secondary Outcome: Change in Antibody Titers
Description: Change in antibody titers 1 month post-dose 3 of vaccine. For each vaccine component, the geometric mean titers (GMT) and the corresponding 95% confidence intervals (CI) were calculated for antibody titers at each time-point (Day 1 and Month 7). For each participant, the difference in antibody titers between these 2 time-points (titers at Month 7 minus titers at Day 1) was calculated. The mean of antibody titer change and its 95% CI were calculated. Immune response was measured with a multiplex competitive Luminex immunoassay (anti-HPV-6, -11, -16, and -18 chemiluminescence immunoassay analyzer (cLIA); Merck) at Pharmaceutical Product Development (PPD). Briefly, this assay simultaneously quantitates neutralizing antibodies to HPV 6, 11, 16, and 18 in 50 μL of serum. mMU/ml is an arbitrary unit of measure derived after comparing relative inhibition of mAb-PE binding to a pooled standard reference serum using a four-parameter logistic curve fit and correcting for dilution.
Time Frame: Points: Day 1 and Month 7
Population: Participants who had specimens contributing to both Day 1 and Month 7 serum HPV antibody evaluations.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL (geometric mean titer)
Groups:
- Gardasil Vaccine - Day 1; Gardasil Vaccine - Month 7: Vaccine Administration: A total of 3 injections (shots) at 3 separate visits.
  Gardasil: The First Shot: Given on the day participants joined the study (Visit 1). The Second Shot: Given about 2 months later (Visit 2). The Third Shot: Given about 6 months after the first (Visit 3).
Arm/Group | Gardasil Vaccine - Day 1 | Gardasil Vaccine - Month 7
Number analyzed (Participants) | 145 | 145
mMU/mL (geometric mean titer)
  HPV 6 | 29.8 [1.4 to 45.9] | 419.5 [363.4 to 484.3]
  HPV 11 | 40.1 [11.1 to 144.5] | 516.6 [454.7 to 586.8]
  HPV 16 | 40.1 [21.4 to 75.1] | 2228.6 [2003.8 to 2478.5]
  HPV 18 | 16.2 [11.8 to 22.2] | 300.0 [259.3 to 347.2]

ADVERSE EVENTS:
Time Frame: 2 years, 3 months
Description: Participants were asked to complete a vaccine report card to document any adverse events for 14 days following each of three doses of vaccine. Trial participants were provided thermometers to record their temperatures each day for five days following each dose of received vaccine.
Arm/Group | Gardasil Vaccine
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 38/150
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gardasil Vaccine (N=150)
Injection site reaction (General disorders) | 19 (29)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (12)
Headache (Nervous system disorders) | 14 (15)

LIMITATIONS AND CAVEATS:
Participants were followed for just 7 months post-dose one of the vaccine; therefore, investigators were unable to assess the durability of the vaccine response in men vaccinated at an older age.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes